CLINICAL TRIAL: NCT05769257
Title: A Phase 2 Multi-Center Safety and Feasibility Study of IS-001 Injection in Patients Undergoing Robotic-Assisted Colorectal Surgery Using the da Vinci® Surgical System With Firefly® Fluorescent Imaging
Brief Title: A Safety and Feasibility Study of IS-001 Injection in Patients Undergoing Robotic Colorectal Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ISI-124804-CR-2
Record Dates: First submitted 2023-01-31; First posted 2023-03-15 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Ureter Injury
MeSH Terms: interventions — IS 001

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Single Arm Safety and Feasibility Study of IS-001 with 20 mg in Multiple Injections
  Interventions: Drug: IS-001

INTERVENTIONS:
Drug: IS-001 — Intravenous injection of IS-001 investigational drug

SUMMARY:
This study evaluates the safety and feasibility of intravenous injection of IS-001 to aid in intraoperative ureter structure delineation

DETAILED DESCRIPTION:
Injury to the ureter, the duct by which urine passes from the kidney into the bladder, is a well-known and serious complication of pelvic and abdominal surgery that frequently goes unrecognized intraoperatively. This study seeks to evaluate the safety and feasibility of intravenous IS-001 injection to improve surgeon ureter visualization during robotic-assisted surgery with the da Vinci® Surgical System and Firefly® imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between the ages of 18 and 75, inclusive
2. Subject is scheduled to undergo robotic-assisted rectal, sigmoid, or left colon resection surgery using the da Vinci® X/Xi Surgical System with Firefly® Fluorescent Imaging

Exclusion Criteria:

1. Subject is pregnant or nursing
2. Subject has known hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
3. Subject has any of the following screening laboratory values:

   1. eGFR < 60 mL/min/1.73 m^2
   2. Aspartate aminotransferase (AST) or serum glutamic oxaloacetic transaminase ≥ 2.5 × ULN
   3. Alanine aminotransferase (ALT) or serum glutamic pyruvic transaminase ≥ 2.5 × ULN
4. Subject is already enrolled in another investigational drug or device study receiving therapeutic agents within the past 6 months
5. Subject has any other condition or personal circumstance that, in the judgment of the Investigator, might interfere with the collection of complete quality data or represents an unacceptable safety profile
6. Subjects with known or suspected hypersensitivity to indocyanine green (ICG) or any components of the formulation used.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Evaluate ureter visualization by Independent Reader | 10 minutes after first IS-001 injection during surgery
  Independent reader assessment of ureter visibility of a 5 second video segment of the surgical field in both Firefly® and standard white light comparator mode on a Five-point rating scale where 1 = Not Visible, 1 = Questionably Visible, 3 = Low Visibility, 4 = Visible, 5 = Clearly Visible
Evaluate ureter visualization by Independent Reader | 30 minutes after first IS-001 injection during surgery
  Independent reader assessment of ureter visibility of a 5 second video segment of the surgical field in both Firefly® and standard white light comparator mode on a Five-point rating scale where 1 = Not Visible, 1 = Questionably Visible, 3 = Low Visibility, 4 = Visible, 5 = Clearly Visible
Evaluate ureter visualization by Independent Reader | 45 minutes after first IS-001 injection during surgery
  Independent reader assessment of ureter visibility of a 5 second video segment of the surgical field in both Firefly® and standard white light comparator mode on a Five-point rating scale where 1 = Not Visible, 1 = Questionably Visible, 3 = Low Visibility, 4 = Visible, 5 = Clearly Visible
Evaluate ureter visualization by Independent Reader | 10 minutes after second IS-001 injection during surgery
  Independent reader assessment of ureter visibility of a 5 second video segment of the surgical field in both Firefly® and standard white light comparator mode on a Five-point rating scale where 1 = Not Visible, 1 = Questionably Visible, 3 = Low Visibility, 4 = Visible, 5 = Clearly Visible
Evaluate ureter visualization by Independent Reader | 30 minutes after second IS-001 injection during surgery
  Independent reader assessment of ureter visibility of a 5 second video segment of the surgical field in both Firefly® and standard white light comparator mode on a Five-point rating scale where 1 = Not Visible, 1 = Questionably Visible, 3 = Low Visibility, 4 = Visible, 5 = Clearly Visible
Evaluate ureter visualization by Independent Reader | 45 minutes after second IS-001 injection during surgery
  Independent reader assessment of ureter visibility of a 5 second video segment of the surgical field in both Firefly® and standard white light comparator mode on a Five-point rating scale where 1 = Not Visible, 1 = Questionably Visible, 3 = Low Visibility, 4 = Visible, 5 = Clearly Visible

SECONDARY OUTCOMES:
Evaluate ureter visualization by Intra-operative surgeon | 10 minutes after first IS-001 injection during surgery
  Intra-operative surgeon assessment of ureter visibility in both Firefly® and standard white light comparator mode on a Five-point rating scale where 1 = Not Visible, 1 = Questionably Visible, 3 = Low Visibility, 4 = Visible, 5 = Clearly Visible
Evaluate ureter visualization by Intra-operative surgeon | 30 minutes after first IS-001 injection during surgery
  Intra-operative surgeon assessment of ureter visibility in both Firefly® and standard white light comparator mode on a Five-point rating scale where 1 = Not Visible, 1 = Questionably Visible, 3 = Low Visibility, 4 = Visible, 5 = Clearly Visible
Evaluate ureter visualization by Intra-operative surgeon | 45 minutes after first IS-001 injection during surgery
  Intra-operative surgeon assessment of ureter visibility in both Firefly® and standard white light comparator mode on a Five-point rating scale where 1 = Not Visible, 1 = Questionably Visible, 3 = Low Visibility, 4 = Visible, 5 = Clearly Visible
Evaluate ureter visualization by Intra-operative surgeon | 10 minutes after second IS-001 injection during surgery
  Intra-operative surgeon assessment of ureter visibility in both Firefly® and standard white light comparator mode on a Five-point rating scale where 1 = Not Visible, 1 = Questionably Visible, 3 = Low Visibility, 4 = Visible, 5 = Clearly Visible
Evaluate ureter visualization by Intra-operative surgeon | 30 minutes after second IS-001 injection during surgery
  Intra-operative surgeon assessment of ureter visibility in both Firefly® and standard white light comparator mode on a Five-point rating scale where 1 = Not Visible, 1 = Questionably Visible, 3 = Low Visibility, 4 = Visible, 5 = Clearly Visible
Evaluate ureter visualization by Intra-operative surgeon | 45 minutes after second IS-001 injection during surgery
  Intra-operative surgeon assessment of ureter visibility in both Firefly® and standard white light comparator mode on a Five-point rating scale where 1 = Not Visible, 1 = Questionably Visible, 3 = Low Visibility, 4 = Visible, 5 = Clearly Visible
Ureter Delineation Efficacy as Length of Line Drawn | 10 minutes after first IS-001 injection during surgery
  Independent reader assessment of ureter delineation on a still frame of the surgical field in both Firefly® and standard white light comparator mode. Length of line drawn on still frame where ureter is visible to independent reader is compared between imaging conditions.
Ureter Delineation Efficacy as Length of Line Drawn | 30 minutes after first IS-001 injection during surgery
  Independent reader assessment of ureter delineation on a still frame of the surgical field in both Firefly® and standard white light comparator mode. Length of line drawn on still frame where ureter is visible to independent reader is compared between imaging conditions.
Ureter Delineation Efficacy as Length of Line Drawn | 45 minutes after first IS-001 injection during surgery
  Independent reader assessment of ureter delineation on a still frame of the surgical field in both Firefly® and standard white light comparator mode. Length of line drawn on still frame where ureter is visible to independent reader is compared between imaging conditions.
Ureter Delineation Efficacy as Length of Line Drawn | 10 minutes after second IS-001 injection during surgery
  Independent reader assessment of ureter delineation on a still frame of the surgical field in both Firefly® and standard white light comparator mode. Length of line drawn on still frame where ureter is visible to independent reader is compared between imaging conditions.
Ureter Delineation Efficacy as Length of Line Drawn | 30 minutes after second IS-001 injection during surgery
  Independent reader assessment of ureter delineation on a still frame of the surgical field in both Firefly® and standard white light comparator mode. Length of line drawn on still frame where ureter is visible to independent reader is compared between imaging conditions.
Ureter Delineation Efficacy as Length of Line Drawn | 45 minutes after second IS-001 injection during surgery
  Independent reader assessment of ureter delineation on a still frame of the surgical field in both Firefly® and standard white light comparator mode. Length of line drawn on still frame where ureter is visible to independent reader is compared between imaging conditions.
Evaluate fluorescent intensity of ureter by signal to background analysis | 10 minutes after first IS-001 injection during surgery
  Fluorescent intensity of ureter evaluated as signal to background
Evaluate fluorescent intensity of ureter by signal to background analysis | 30 minutes after first IS-001 injection during surgery
  Fluorescent intensity of ureter evaluated as signal to background
Evaluate fluorescent intensity of ureter by signal to background analysis | 45 minutes after first IS-001 injection during surgery
  Fluorescent intensity of ureter evaluated as signal to background
Evaluate fluorescent intensity of ureter by signal to background analysis | 10 minutes after second IS-001 injection during surgery
  Fluorescent intensity of ureter evaluated as signal to background
Evaluate fluorescent intensity of ureter by signal to background analysis | 30 minutes after second IS-001 injection during surgery
  Fluorescent intensity of ureter evaluated as signal to background
Evaluate fluorescent intensity of ureter by signal to background analysis | 45 minutes after second IS-001 injection during surgery
  Fluorescent intensity of ureter evaluated as signal to background
Safety 12-Lead EKG Change from Baseline | 6 hours after first IS-001 injection post surgery
  12-Lead EKG change from baseline in QTc
Incidence of abnormal blood work in tests results | Before same-day discharge or 24 hours after first IS-001 injection post surgery
  Safety hematology complete blood count laboratory assessments Change from Baseline
Incidence of abnormal blood work in tests results | Before same-day discharge or 24 hours after first IS-001 injection post surgery
  Safety hematology comprehensive metabolic panel laboratory assessments Change from Baseline
Incidence of abnormal blood work in tests results | 14 days post surgery
  Safety hematology complete blood count laboratory assessments Change from Baseline
Incidence of abnormal blood work in tests results | 14 days post surgery
  Safety hematology comprehensive metabolic panel laboratory assessments Change from Baseline
Incidence of abnormal urinalysis results | 14 days post surgery
  Routine urinalysis laboratory assessment change from baseline
Safety Adverse Events Monitoring | 14 days post surgery
  Drug related adverse events monitoring through 14-days

CONTACTS AND LOCATIONS:
Overall Officials: Thiru Lakshman, MD, Principal Investigator — St. David's North Austin Medical Center; Laila Rashidi, MD, Principal Investigator — MultiCare Tacoma General Hospital
Locations (2):
- United States (2):
  - St. David's North Austin Medical Center, Austin, Texas
  - MultiCare Tacoma General Hospital, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No